CLINICAL TRIAL: NCT06363591
Title: Wise vs Wide: A National, Multicenter, Prospective, Randomized and Controlled, Parallel Group, Non-inferiority Study to Compare Single- vs Two-staged Excisions of Thin Melanoma
Brief Title: WoW - Single- vs Two-staged Excisions of Thin Melanoma
Acronym: WoW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Region Stockholm (Other Government); Region Skane (Other); Region Västerbotten (Other Government); Region Örebro County (Other); Blekinge County Council Hospital (Other); Region Östergötland (Other); Dalarna County Council, Sweden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WoW - Wise or wide
Record Dates: First submitted 2024-03-28; First posted 2024-04-12 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-01

CONDITIONS: Melanoma
Keywords: Melanoma; Surgery; Wide local excision; Recurrence; Metastasis; Death
MeSH Terms: conditions — Melanoma; Recurrence; Neoplasm Metastasis; Death | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Patients with thin (≤1.0 mm) invasive melanomas excised with a histopathological margin ≥1.5 mm will be offered to participate following informed consent and randomization (1:1) to either:
  1. Standard treatment with a WLE of the diagnostic excision scar with a lateral clinical surgical margin of 10 mm and a deep clinical surgical margin down to the muscular fascia as recommended by the Swedish national guidelines.
     or
  2. Experimental treatment with no WLE.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wide - With wide local excision - Control group (Other): Standard treatment with a wide local excision (i.e. reexcision of the diagnostic excision scar with a lateral clinical surgical margin of 10 mm and a deep clinical surgical margin down to the muscular fascia as recommended by the Swedish national guidelines).
  Interventions: Procedure: Surgery
- Wise - Without wide local excision - Experimental group (Experimental): No wide local excision.
  Interventions: Other: No Surgery

INTERVENTIONS:
Procedure: Surgery — Wise or wide excision
  Arms: Wide - With wide local excision - Control group
Other: No Surgery — No wide local excision
  Arms: Wise - Without wide local excision - Experimental group

SUMMARY:
The overall aim of this national, multicenter, prospective, randomized, and controlled study is to enhance the management of patients with thin melanoma (≤1 mm Breslow thickness). The investigators hypothesize that wide local excisions (WLEs) following complete excision of thin melanoma do not affect the risk of recurrence, defined as the occurrence of local, regional, distant disease, or melanoma-specific death during a 5- to 10-year follow-up period.

DETAILED DESCRIPTION:
Melanoma is one of the most common forms of skin cancer and has become the third most common type of cancer among men and the fourth most common among women in Sweden.

The mortality associated with melanoma is strongly linked to the thickness of the original tumor. Thicker tumors generally have a worse prognosis compared to thinner tumors. In melanoma in situ (MIS), the tumor is confined to the epidermis and cannot spread. In invasive melanoma, the tumor has grown into the dermis. The thickness of these invasive melanomas is measured using the "Breslow thickness." Thinner invasive melanomas with a Breslow thickness of ≤1.0 mm constitute the majority of cases in Sweden and have an excellent prognosis with a 10-year disease-specific survival rate of 97%.

Melanoma represents a significant economic burden with increasing healthcare costs. Early detection and cost-effective treatment strategies are therefore important to improve prognosis, reduce costs, and avoid unnecessary overtreatment.

Surgical methods for treating melanoma vary depending on the thickness of the tumor. Traditionally, a two-step procedure has been used. Initially, a diagnostic excision (surgery to remove the tumor) with a narrow clinical margin is performed. Once melanoma is confirmed, a second wide local excision (WLE) is performed around the surgical scar with a 1-2 cm clinical margin depending on the exact Breslow thickness. This method has evolved over time, and narrower clinical margins are now used in the WLE than previously. However, researchers have begun to question whether a WLE is necessary at all for thin melanomas if the tumor is completely removed during the initial diagnostic excision.

Researchers are now exploring a more personalized treatment strategy that considers histopathological margins instead of a standardized clinical margin. For well-defined melanomas, a clinical margin of 3-5 mm may be sufficient to ensure that the melanoma is removed with an acceptable histopathological margin (≥1.5 mm). The hypothesis is that this margin may be adequate and that the WLE does not reduce the risk of local, regional or distant disease nor melanoma-specific death. If the hypothesis is proven, unnecessary surgery, patient suffering, risk of complications, resource utilization, and healthcare costs could be reduced.

The investigators now want to investigate whether there is a difference in the risk of recurrence, spread, and/or death for patients with thin melanomas (≤1mm Breslow thickness) treated with only one excision compared to the current standard of two excisions.

ELIGIBILITY:
Inclusion Criteria:

Patients need to fulfill all criteria listed below:

* Has recently been diagnosed with a primary invasive cutaneous melanoma of Breslow thickness ≤1.0 mm (pT1) as determined by a diagnostic excision with subsequent histopathological analysis that:

  1. Is located on a body location in which a WLE with a 10-mm clinical margin is feasible and would have been planned according to current standard of care.
  2. Had histopathologically verified free margins of at least 1.5 mm.
* Is 18 years or older at time of consent.
* Is able to give informed consent and comply with the treatment protocol and follow-up plan.
* Has a life expectancy of ≥5 years from the time of diagnosis.

Exclusion Criteria:

If any of the listed criteria below are present, the patient is ineligible for study participation.

The study lesion:

* was partially biopsied prior to the diagnostic excision.
* was diagnostically excised with a clinical margin >5 mm.
* was a melanoma of desmoplastic or lentiginous (i.e. lentigo maligna or acral lentiginous) subtype.
* was located on digits in which amputation is necessary.

The patient:

* had a previous or concurrent MIS or invasive melanoma (cutaneous or non-cutaneous).
* had physical, clinical, radiographic or pathologic evidence of microsatellite, satellite, in-transit, regional or distant metastatic melanoma.
* had a previous or intercurrent treated solid tumor or hematologic malignancy during the past 5 years except cutaneous squamous cell carcinoma or basal cell carcinoma.
* has planned adjuvant radiotherapy to the primary melanoma site after WLE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2486 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2039-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate at 5 years. | 5 years
  Recurrence is defined as any presence of local/regional/distant disease or melanoma-specific death.

SECONDARY OUTCOMES:
Recurrence rate at 10 years. | 10 years
  Recurrence is defined as any presence of local/regional/distant disease or melanoma-specific death.

OTHER OUTCOMES:
Postoperative complications | 3 months
  Determine the frequency of postoperative complications in both treatment groups.
Scar length, width and quality | 1 year
  Measurement of the scar length and width as well as the scar quality assessed by both patient and clinician (measured with the Patient and Observer Scar Assessment Scale, POSAS). The POSAS consists of two subscales: the Patient Scale and the Observer Scale, each ranging from 6 to 60, where a lower score indicates a better scar outcome.
Scar length, width and quality | 3 years
  Measurement of the scar length and width as well as the scar quality assessed by both patient and clinician (measured with the Patient and Observer Scar Assessment Scale, POSAS). The POSAS consists of two subscales: the Patient Scale and the Observer Scale, each ranging from 6 to 60, where a lower score indicates a better scar outcome.
Patient satisfaction | 3 months
  The Functional Assessment of Chronic Illness Therapy - Treatment Satisfaction - Patient Satisfaction questionnaire (FACIT-TS-PS) is to be completed electronically or in clinic. The FACIT-TS-PS assesses patient satisfaction with treatment, with total scores ranging from 0 to 36, where higher scores indicate greater satisfaction with treatment.
Patient satisfaction | 1 year
  The Functional Assessment of Chronic Illness Therapy - Treatment Satisfaction - Patient Satisfaction questionnaire (FACIT-TS-PS) is to be completed electronically or in clinic. The FACIT-TS-PS assesses patient satisfaction with treatment, with total scores ranging from 0 to 36, where higher scores indicate greater satisfaction with treatment.
Patient satisfaction | 2 years
  The Functional Assessment of Chronic Illness Therapy - Treatment Satisfaction - Patient Satisfaction questionnaire (FACIT-TS-PS) is to be completed electronically or in clinic. The FACIT-TS-PS assesses patient satisfaction with treatment, with total scores ranging from 0 to 36, where higher scores indicate greater satisfaction with treatment.
Patients' quality of life | 3 months
  The Quality of Life (QoL) questionnaire Functional Assessment of Cancer Therapy - Melanoma (FACT-M) is to be completed electronically or in clinic. The FACT-M assesses quality of life in melanoma patients, with total scores ranging from 0 to 172, where higher scores indicate better quality of life.
Patients' quality of life | 1 year
  The Quality of Life (QoL) questionnaire Functional Assessment of Cancer Therapy - Melanoma (FACT-M) is to be completed electronically or in clinic. The FACT-M assesses quality of life in melanoma patients, with total scores ranging from 0 to 172, where higher scores indicate better quality of life.
Patients' quality of life | 2 years
  The Quality of Life (QoL) questionnaire Functional Assessment of Cancer Therapy - Melanoma (FACT-M) is to be completed electronically or in clinic. The FACT-M assesses quality of life in melanoma patients, with total scores ranging from 0 to 172, where higher scores indicate better quality of life.
All-cause mortality | 5 years
  Overall all-cause mortality incidence in both treatment groups.
All-cause mortality | 10 years
  Overall all-cause mortality incidence in both treatment groups.
Direct and indirect costs per patient | 5 years
  Calculate and compare costs per patient in the experimental and control groups.
Biomarkers | 10 years
  Differences in biomarkers of recurrent and non-recurrent melanomas.

CONTACTS AND LOCATIONS:
Overall Officials: John Paoli, Professor, Principal Investigator — Dept. of Dermatology and Venereology, Sahlgrenska Academy, University of Gothenburg, Sweden
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available 6 months after publication of study results (start date) and 1 year after this (end date).
Access Criteria: Data will be shared upon reasonable request and accessed by contacting john.paoli@gu.se.
URL: https://www.gu.se/en/about/find-staff/johnpaoli

REFERENCES:
- [Derived] Wennberg E, Claeson M, Olofsson Bagge R, Polesie S, Paoli J. Wise or wide (WoW) study protocol: a national, multicentre, prospective, randomised and controlled, parallel group, non-inferiority study to compare single-staged versus two-staged excisions of thin invasive (</=1.0 mm) melanoma. BMJ Open. 2025 Apr 2;15(4):e094544. doi: 10.1136/bmjopen-2024-094544. PMID 40180392